CLINICAL TRIAL: NCT00003942
Title: A Phase I/II Study of the Safety and Feasibility of REVM10 or REVM10/ANTISENSE POL 1 Transduced Hematopoietic Stem Cells (HSC) in HIV-1 Related Non-Hodgkin's Lymphoma Patients Already Being Treated With High Dose Chemotherapy and Peripheral Blood Stem Cell Support
Brief Title: Gene Therapy, Chemotherapy, and Peripheral Stem Cell Transplantation in Treating Patients With HIV-Related Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Systemix (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067135; SYSTEMIX-105; UCLA-HSPC-980303601D; NCI-G99-1549
Record Dates: First submitted 1999-11-01; First posted 2004-07-26 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2000-08

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: RevM10 gene
Biological: RevM10/polAS gene
Procedure: in vitro-treated peripheral blood stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Inserting the gene for RevM10 into a person's peripheral stem cells may improve the body's ability to fight cancer or make the cancer more sensitive to chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of RevM10-treated stem cells plus chemotherapy and peripheral stem cell transplantation in treating patients who have HIV-related non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of infusion of RevM10 or RevM10/polAS transduced hematopoietic stem cells (HSC) in addition to high dose chemotherapy and standard peripheral blood stem cell support in patients with HIV-1 related non-Hodgkin's lymphoma. II. Determine gene marking of lymphocytes and myeloid cells in peripheral blood, bone marrow, and/or lymph nodes after infusion of RevM10-HSC or RevM10/polAS-HSC in these patients. III. Determine the antiretroviral effect of this treatment in these patients.

OUTLINE: This is a multicenter study. Patients receive mobilization therapy and undergo leukapheresis according to a standard protocol. High dose chemotherapy is administered on days -7 to -1, also according to a standard protocol. On day 0, autologous hematopoietic stem cells transduced with genes RevM10 or RevM10/polAS are infused. Unmodified autologous peripheral blood stem cells are reinfused on day 1. Patients are followed daily for 2 weeks, weekly for 2 weeks, monthly for 1 year, then annually thereafter.

PROJECTED ACCRUAL: Approximately 15 patients will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: HIV-1 infection documented by ELISA and Western blot Histologically proven non-Hodgkin's lymphoma showing at least partial response to standard chemotherapy regimen Poor prognosis in first chemotherapy induced remission Increased LDH AND/OR Stage III or IV AND/OR Reduced performance status (ECOG 2 or worse) OR Response but no complete remission following four courses of standard chemotherapy OR Responding relapse after primary therapy No primary CNS lymphoma No uncontrolled meningeal lymphoma at mobilization

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: See Disease Characteristics Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 CD4 count at least 100/mm3 Hepatic: Bilirubin less than 2 mg/dL (unless taking indinavir) SGOT and SGPT less than 2 times normal No hepatitis Renal: Creatinine less than 2.0 mg/dL Pulmonary: DLCO greater than 60% Other: Not pregnant or nursing Fertile patients must use effective contraception No active Mycobacterium avium-intracellulare infection or CMV disease No cerebral toxoplasmosis or cryptococcal meningitis At least 6 months since prior alcohol or substance abuse At least 1 year since CNS disease or seizures No other medical condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No concurrent chemotherapy for Kaposi's sarcoma Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 30 days since prior treatment for serious opportunistic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 1998-11

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Martin, MD, Study Chair — Systemix
Locations (6):
- United States (6):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Division of Oncology, Palo Alto, California
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska